CLINICAL TRIAL: NCT04843475
Title: Study of Pulmonary Hypertension in Patients With Chronic Myeloproliferative Disorders at Sohag University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Hamdy Ahmed, assistant lecturer, Sohag University
Other Study IDs: Soh-Med-21-04-15
Record Dates: First submitted 2021-04-12; First posted 2021-04-13 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Chronic Myeloproliferative Disorders
MeSH Terms: conditions — Myeloproliferative Disorders | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MPNs patients who have echocardiographic probability of PH.
  Interventions: Diagnostic Test: Echocardiography
- MPNs patients who do not have echocardiographic probability of PH
  Interventions: Diagnostic Test: Echocardiography

INTERVENTIONS:
Diagnostic Test: Echocardiography — Trans-thoracic Echocardiography

SUMMARY:
Pulmonary hypertension (PH) is a complex condition that may be related to many clinical conditions. It is a serious disorder with a high morbidity and mortality rates. PH is classified into five groups according to clinical characteristics, pathological findings, hemodynamic characteristics and treatment response (Galie N, et al., 2016). These five groups include pulmonary arterial hypertension, PH due to left sided heart disease, PH due to lung disease and/or hypoxia, chronic thromboembolic pulmonary hypertension, or other pulmonary arterial obstruction and PH with unclear and/or multifactorial mechanisms (Simonneau G, et al., 2013).

PH is a major complication of several hematologic disorders including myeloproliferative neoplasms (MPNs). MPNs are a group of diseases characterized by uncontrolled proliferation of at least one myeloid series due to an abnormal hematopoietic cell clone. There are different types of MPNs including polycythemia vera (PV), essential thrombocythemia (ET), primary myelofibrosis (PMF) & chronic myeloid leukemia ( CML). Myeloproliferative neoplasms (MPNs) are included in group 5 PH (Arber DA, et al., 2016).

This study will analyze the clinical and laboratory data of MPNs patients and correlate them with development of PH in these patients aiming to identify parameters that can predict PH in MPNs patients and thus, identifying MPNs patients at highest risk for PH who require close monitoring & screening for PH hoping that early detection and management of PH in MPNs patients can improve morbidity, prognosis and survival in those patients

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old.
* Patients diagnosed with polycythemia vera, essential thrombocythemia, primary myelofibrosis and chronic myeloid leukemia according to the 2016 WHO classification and attended the outpatient Hematology Clinic at Sohag University Hospital.

Exclusion Criteria:

* Patients less than 18 years old.
* Patients with pre-existing pulmonary hypertension from any other cause.
* Patients with left sided heart disease e.g. left sided heart failure, left sided valvular diseases, cardiomyopathies, left ventricular systolic or diastolic dysfunction.
* Patients with chronic lung disease e.g. COPD & interstitial lung disease.
* Patients with chronic kidney disease.
* Patients with connective tissue diseases.
* Patients with congenital heart diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The outpatient Hematology Clinic at Sohag University Hospital.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of pulmonary hypertension in chronic myeloproliferative disorders patients | 2 years
  Prevalence of pulmonary hypertension in chronic myeloproliferative disorders patients

SECONDARY OUTCOMES:
Identification of independent different predictors of pulmonary hypertension in chronic myeloproliferative disorders patients | 2 years
  Identification of independent different predictors of pulmonary hypertension in chronic myeloproliferative disorders patients

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Galie N, Humbert M, Vachiery JL, Gibbs S, Lang I, Torbicki A, Simonneau G, Peacock A, Vonk Noordegraaf A, Beghetti M, Ghofrani A, Gomez Sanchez MA, Hansmann G, Klepetko W, Lancellotti P, Matucci M, McDonagh T, Pierard LA, Trindade PT, Zompatori M, Hoeper M; ESC Scientific Document Group. 2015 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension: The Joint Task Force for the Diagnosis and Treatment of Pulmonary Hypertension of the European Society of Cardiology (ESC) and the European Respiratory Society (ERS): Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC), International Society for Heart and Lung Transplantation (ISHLT). Eur Heart J. 2016 Jan 1;37(1):67-119. doi: 10.1093/eurheartj/ehv317. Epub 2015 Aug 29. No abstract available. PMID 26320113
- [Background] Yaylali YT, Yilmaz S, Akgun-Cagliyan G, Kilic O, Kaya E, Senol H, Ozen F. Association of Disease Subtype and Duration with Echocardiographic Evidence of Pulmonary Hypertension in Myeloproliferative Neoplasm. Med Princ Pract. 2020;29(5):486-491. doi: 10.1159/000506596. Epub 2020 Feb 19. PMID 32069470
- [Background] Lopez-Mattei J, Verstovsek S, Fellman B, Iliescu C, Bhatti K, Hassan SA, Kim P, Gray BA, Palaskas NL, Grosu HB, Mamas MA, Faiz SA. Prevalence of pulmonary hypertension in myelofibrosis. Ann Hematol. 2020 Apr;99(4):781-789. doi: 10.1007/s00277-020-03962-2. Epub 2020 Feb 19. PMID 32076825